CLINICAL TRIAL: NCT06178406
Title: Brain Structural and Functional Connectivity Changes in the Period of Dysmenorrhea: a Prospective Functional Magnetic Resonance Imaging Study
Brief Title: Brain Structural and Functional Connectivity Changes in the Period of Dysmenorrhea: a Prospective fMRI Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20230284-R
Record Dates: First submitted 2023-09-04; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Dysmenorrhea
Keywords: dysmenorrhea, magnetic resonance imaging
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dysmenorrhea
  Interventions: Behavioral: dysmenorrhea
- female healthy controls

INTERVENTIONS:
Behavioral: dysmenorrhea — Dysmenorrhea, defined as painful menstrual cramps of uterine origin, is the most common gynecological condition among women of reproductive age.
  Groups: dysmenorrhea

SUMMARY:
Observational prospective study with an analysis of the changes in brain structure and related functional connectivity in women with dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea is a common gynecological disease and chronic pain disorder.Understanding the neural mechanisms of dysmenorrhea and the brain changes affecting pain factors is important for finding dysmenorrhea treatment methods. The emergence and progress of non-invasive neuroimaging technology can help us better understand pain at the neural level. Recent developments in identifying brain-based biomarkers of pain through advances in advanced imaging can provide some foundations for predicting and detecting pain. Twenty patients with dysmenorrhea and twenty matched female healthy controls were recruited from our hospital. All participants underwent the head magnetic resonance imaging scans to calculate grey matter volume and Diffusion Tensor Imaging parameters. Questionnaire assessment was also conducted.

ELIGIBILITY:
Inclusion Criteria:

* Right-handedness, as confirmed by the Edinburgh Handedness Inventory
* A regular menstrual cycle of approximately 21 to 35 days
* A history of menstrual pain longer than 6 months
* Not taking any medication or using other methods to treat dysmenorrhea in the past month
* Score of >= 40mm on the VAS (visual analogue scale) in recent three menstrual cycles

Exclusion Criteria:

* Any psychiatric or neurological disorders, particularly premenstrual dysphoric disorder
* Using oral contraceptives, hormonal supplements, or any central-acting medication (eg, opioid, antiepileptics) within 6 months before the study
* Having a metal or pacemaker implant, claustrophobia, or any contraindications to MR
* Head injury with loss of consciousness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the patients with dysmenorrhea underwent pelvic ultrasonography to identify the cause of dysmenorrhea. The study will be conducted in accordance with the Declaration of Helsinki and approved by the Institutional Review Board of Women's Hospital School of Medicine Zhejiang University. All participants will give their written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The functional connectivity of functional magnetic resonance imaging | 1 month
  Functional magnetic resonance imaging (fMRI)-based functional connectivity (FC) commonly characterizes the functional connections in the brain.

SECONDARY OUTCOMES:
Grey Matter volume | 1 month
  the grey matter volume is defined as the amount of grey matter that lies between the grey-white interface and the pia mater.